CLINICAL TRIAL: NCT03094832
Title: A Phase 1/2 Study of ARQ 092 (Miransertib) in Subjects With PIK3CA-related Overgrowth Spectrum and Proteus Syndrome
Brief Title: Study of Miransertib (MK-7075) in Participants With PIK3CA-related Overgrowth Spectrum and Proteus Syndrome (MOSAIC) (MK-7075-002)
Acronym: MOSAIC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Early termination due to business reasons
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7075-002; MOSAIC (Other: ArQule); ARQ 092-103 (Other: ArQule); MK-7075-002 (Other: Merck); 2016-000558-37 (EudraCT Number)
Expanded Access: NCT03317366 (No longer available)
Record Dates: First submitted 2017-03-17; First posted 2017-03-29 (Actual); Results first posted 2023-03-31 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: PIK3CA-Related Overgrowth Spectrum (PROS)/Proteus Syndrome
Keywords: ARQ 092; ArQule; AKT; PIK3CA; Overgrowth; Congenital malformations; Miransertib; MOSAIC
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies; Congenital Abnormalities | interventions — Miransertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: Miransertib PROS/PS (Experimental): During Cycles 1-3, participants with either PROS (phosphatidylinositol- 4,5-bisphosphate 3-kinase, catalytic subunit alpha [PIK3CA]-related Overgrowth Spectrum) or PS (Proteus syndrome) received miransertib 15 mg/m^2 once daily (QD) (each cycle length = 28 days). From Cycles 4-48 or until disease progression, unacceptable toxicity, or discontinuation, participants received miransertib dose titrated to 25 mg/m^2 and then titrated to 35 mg/m^2 orally QD at the investigator's discretion.
  Interventions: Drug: Miransertib
- Part B: Miransertib PROS (Cohort 1) (Experimental): During Cycles 1-3, participants with PROS who have a measurable lesion by volumetric magnetic resonance imaging (MRI) received miransertib 15 mg/m^2 QD (each cycle length = 28 days). From cycles 4-48 or until disease progression, unacceptable toxicity, or discontinuation, participants received miransertib dose titrated to 25 mg/m^2 orally QD at the investigator's discretion.
  Interventions: Drug: Miransertib
- Part B: Miransertib PS (Cohort 2) (Experimental): During Cycles 1-3, participants with PS who have a measurable lesion by standardized digital photography received miransertib 15 mg/m^2 QD (each cycle length = 28 days). From cycles 4-48 or until disease progression, unacceptable toxicity, or discontinuation, participants received miransertib dose titrated to 25 mg/m^2 orally QD at the investigator's discretion.
  Interventions: Drug: Miransertib
- Part B: Miransertib PROS/PS (Cohort 3) (Experimental): During Cycles 1-3, participants with PROS or PS who do not meet all the eligibility criteria for Cohorts 1 or 2 received miransertib 15 mg/m^2 QD (each cycle length = 28 days). From cycles 4-48 or until disease progression, unacceptable toxicity, or discontinuation, participants received miransertib dose titrated to 25 mg/m^2 orally QD at the investigator's discretion.
  Interventions: Drug: Miransertib
- Part B: Miransertib Compassionate Use/Expanded Access (Cohort 4) (Experimental): During cycles 1-48 (each cycle length = 28 days) or until disease progression, unacceptable toxicity, or discontinuation, participants previously treated with miransertib or currently receiving miransertib under Compassionate Use/Expanded Access continued to receive the current dose of miransertib (did not exceed 25 mg/m^2).
  Interventions: Drug: Miransertib

INTERVENTIONS:
Drug: Miransertib — Miransertib capsules administered orally at an initial dose of 15 mg/m^2 or 25 mg/m^2 QD and then titrated up to 25 mg/m^2 or 35 mg/m^2 QD at the investigator's discretion.
  Other Names: MK-7075; ARQ 092

SUMMARY:
This is an open label, Phase 1/2 study of oral miransertib (MK-7075) administered to participants at least 2 years of age with phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA)-related Overgrowth Spectrum (PROS) and Proteus Syndrome (PS) (MOSAIC).

DETAILED DESCRIPTION:
The study consists of two parts: Part A and Part B. Part A was closed to enrollment under Amendment 6. As of Amendment 7, the endpoints for Part A and Part B have been combined to assess the safety and tolerability of miransertib in participants with PROS and PS. Previous efficacy and pharmacokinetic (PK) objectives and endpoints have been removed. Amendment 7 will complete the final enrollment into the MOSAIC study and Compassionate Use/Expanded Access Program.

ELIGIBILITY:
Inclusion Criteria:

Part A

* Signed informed consent and, when applicable, signed assent
* Male or female participants ≥ 2 years old with body surface area (BSA) of ≥ 0.33 m^2
* Have a clinical diagnosis of PROS or PS with documented somatic PIK3CA or serine-threonine protein kinase (AKT1) mutations
* Archival or fresh overgrowth tissue sample available to be shipped to Sponsor or designee
* Have poor prognosis, significant morbidity, and/or progressive disease (e.g., worsening of the disease/increase in number or size of the overgrowth lesions in the last 12 months)
* Have measurable disease (at least one overgrowth lesion that can be accurately measured in size by imaging and/or linear or circumference measure)
* Adequate organ function based on screening laboratory values
* If a female is of child-bearing potential, documentation of a negative pregnancy test is required prior to enrollment. Sexually active participants (male and female) must agree to use double-barrier contraceptive measures, oral contraception, or avoidance of intercourse while on study and for up to 90 days after ending treatment
* Ability to complete the Quality of Life (QoL) questionnaires by the participant or his/her caregiver

Part B:

* Signed consent form and when applicable, signed assent
* Archival or fresh overgrowth tissue sample available to be shipped to Sponsor or designee
* Except for Cohort 4, clinically progressive or worsening disease defined as an increase in number or size of the overgrowth lesion(s) in the last 6 months as assessed by the Investigator
* Adequate organ function based on screening laboratory values
* Male or female participants of child-producing potential must agree to use double-barrier contraceptive measures, oral contraception, or avoidance of intercourse during the study and for 90 days after the last dose of miransertib
* Ability to complete the study questionnaires by the participant or his/her caregiver

Cohort 1 (PROS) specific criteria

* Male or female participants ≥ 2 years and ≤30 years of age with BSA of ≥ 0.33 m2
* Have clinical diagnosis of PROS per Diagnostic Criteria for PROS and documented somatic PIK3CA variant
* Have at least one lesion that can be measured by study- standardized volumetric MRI (eligibility to be confirmed by blinded independent central imaging review

  - Cohort 2 (PS) specific criteria
* Male or female participants ≥ 2 years and ≤18 years of age with BSA of ≥ 0.33 m2
* Have clinical diagnosis of PS per Diagnostic Criteria for PS and documented somatic AKT1 variant
* Have at least one plantar cerebriform connective tissue nevus (CCTN) and pre-CCTN lesion that can be measured by standardized photography

  * Cohort 3 specific criteria: Male or female participants ≥2 years old with BSA of ≥ 0.33 m2 and who fail to meet the eligibility criteria for Cohorts 1 or 2
  * Cohort 4 (PROS or PS) specific criteria: participants previously treated with miransertib or currently receiving miransertib under Compassionate Use/Expanded Access. Participants should meet the age criterion by/on the date of the first dose, Cycle 1 Day 1

Exclusion Criteria

Part A:

* History of Type 1 or 2 uncontrolled diabetes mellitus requiring regular medication (other than metformin or other oral hypoglycemic agents) or fasting glucose ≥ 160 mg/dL (if > 12 years old) and ≥ 180 mg/dL (if ≤ 12 years old) at the screening visit
* History of significant cardiac disorders:

  * Myocardial infarction (MI) or congestive heart failure defined as Class II-IV per the New York Heart Association (NYHA) classification within 6 months of the first dose of miransertib (MI occurring > 6 months of the first dose of miransertib will be permitted)
  * Grade 2 (per NCI CTCAE version 4.03) or worse conduction defect (e.g., right or left bundle branch block); left ventricular ejection fraction (LVEF) < 50% assessed by echocardiogram/multigated acquisition (MUGA) scan
* Major surgery, radiotherapy, or immunotherapy within four weeks of the first dose of miransertib
* Any experimental systemic therapy for the purpose of treating PROS or PS (e.g., sirolimus, everolimus, high dose steroids) within two weeks of the first dose of miransertib, except for participants who were previously or are currently treated with miransertib under a Compassionate Use/Expanded Access program
* Intolerance of or severe toxicity attributed to v-Akt murine thymoma viral oncogene homolog (AKT) inhibitors (e.g., miransertib, uprosertib, afuresertib, ipatasertib)
* Concurrent severe uncontrolled illness not related to PROS or PS (ongoing or active infection, known human immunodeficiency virus (HIV) infection, malabsorption syndrome, psychiatric illness/substance abuse/social situation that would limit compliance with study requirements)
* Pregnant or breastfeeding
* Inability to comply with study evaluations or to follow drug administration guidelines

Part B

* History of Type 1 diabetes mellitus or Type 2 uncontrolled diabetes mellitus requiring regular medication (other than metformin or other oral hypoglycemic agents) or fasting glucose ≥ 160 mg/dL (if > 12 years old) and ≥ 180 mg/dL (if ≤ 12 years old) at the screening visit
* History of significant cardiac disorders:

  * Myocardial infarction (MI) or congestive heart failure defined as Class II-IV per the New York Heart Association (NYHA) classification within 6 months of the first dose of miransertib (MI occurring > 6 months of the first dose of miransertib will be permitted)
  * Grade 2 (per current version of National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE]) or worse conduction defect (e.g., right or left bundle branch block)
  * Major surgery or locoregional therapy within four weeks of the first dose of miransertib
* Any experimental systemic therapy for the purposes of treating PROS or PS (e.g., sirolimus, everolimus, high dose steroids) within two weeks of the first dose of miransertib
* Intolerance of or severe toxicity attributed to AKT inhibitors (e.g., miransertib, uprosertib, afuresertib, ipatasertib)
* Concurrent severe uncontrolled illness not related to PROS or PS (e.g. ongoing or active infection, known HIV infection, malabsorption syndrome, psychiatric illness/substance abuse/social situation that would limit compliance with study requirements)
* Pregnant or breastfeeding
* Inability to comply with study evaluations or to follow drug administration guidelines

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (11):
- United States (6):
  - Children's Hospital of Atlanta ( Site 0107), Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago ( Site 0101), Chicago, Illinois
  - Boston Children's Hospital ( Site 0089), Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center ( Site 0102), Cincinnati, Ohio
  - Texas Children's Hospital ( Site 0104), Houston, Texas
  - Seattle Childrens Hospital ( Site 0103), Seattle, Washington
- Hunter Genetics ( Site 0201), Waratah NSW, New South Wales, Australia
- Italy (3):
  - Ospedale Pediatrico Bambino Gesu ( Site 0087), Rome, Roma
  - Universita di Catania ( Site 0088), Catania
  - Fondazione Policlinico Universitario A. Gemelli ( Site 0052), Roma
- Hospital Sant Joan ( Site 0601), Esplugues de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Eng W, Iacobas I, Perkins J, Zampino G, Leoni C, Buonuomo PS, Simonetti A, Goel H, Briones M, Huang M, Goldmacher G, Liaw D, Hammill A. Safety findings from the phase 1/2 MOSAIC study of miransertib for patients with PIK3CA-related overgrowth spectrum or Proteus syndrome. Orphanet J Rare Dis. 2025 Jul 25;20(1):375. doi: 10.1186/s13023-025-03831-z. PMID 40713644
- [Derived] Forde K, Resta N, Ranieri C, Rea D, Kubassova O, Hinton M, Andrews KA, Semple R, Irvine AD, Dvorakova V. Clinical experience with the AKT1 inhibitor miransertib in two children with PIK3CA-related overgrowth syndrome. Orphanet J Rare Dis. 2021 Feb 27;16(1):109. doi: 10.1186/s13023-021-01745-0. PMID 33639990

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 50 participants were enrolled in the study of which 49 participants received at least one dose of treatment and was used for safety analysis.
Groups:
- Part B:Miransertib Compassionate Use/Expanded Access(Cohort 4): During cycles 1-48 (each cycle length = 28 days) or until disease progression, unacceptable toxicity, or discontinuation, participants previously treated with miransertib or currently receiving miransertib under Compassionate Use/Expanded Access continued to receive the current dose of miransertib (did not exceed 25 mg/m^2).
Period: Overall Study
Arm/Group | Part A: Miransertib PROS/PS | Part B: Miransertib PROS (Cohort 1) | Part B: Miransertib PS (Cohort 2) | Part B: Miransertib PROS/PS (Cohort 3) | Part B:Miransertib Compassionate Use/Expanded Access(Cohort 4)
Started | 17 | 22 | 1 | 8 | 2
Treated | 17 | 22 | 1 | 8 | 1
Completed | 2 | 2 | 0 | 0 | 0
Not Completed | 15 | 20 | 1 | 8 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 1 | 0 | 0 | 0 | 0
Not completed — Other | 13 | 20 | 1 | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Miransertib PROS/PS | Part B: Miransertib PROS (Cohort 1) | Part B: Miransertib PS (Cohort 2) | Part B: Miransertib PROS/PS (Cohort 3) | Part B:Miransertib Compassionate Use/Expanded Access(Cohort 4) | Total
Number analyzed (Participants) | 17 | 22 | 1 | 8 | 2 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.2 (9.9) | 9.9 (6.7) | 12.0 (NA) — Standard deviation was not calculatable when n<2. | 12.5 (9.1) | 20.0 (1.4) | 10.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 0 | 3 | 1 | 23
  Male | 8 | 12 | 1 | 5 | 1 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 15 | 20 | 1 | 8 | 2 | 46
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 0 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 5 | 0 | 1 | 0 | 6
  White | 17 | 13 | 1 | 6 | 2 | 39
  More than one race | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product and does not imply any judgment about causality.
Time Frame: Up to approximately 48 months
Population: All participants who have received at least one dose of study treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Miransertib PROS/PS | Part B: Miransertib PROS (Cohort 1) | Part B: Miransertib PS (Cohort 2) | Part B: Miransertib PROS/PS (Cohort 3) | Part B:Miransertib Compassionate Use/Expanded Access(Cohort 4)
Number analyzed (Participants) | 17 | 22 | 1 | 8 | 1
Participants | 17 | 20 | 0 | 6 | 1

2. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: as for outcome 1
Time Frame: Up to approximately 45 months
Population: All participants who have received at least one dose of study treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Miransertib PROS/PS | Part B: Miransertib PROS (Cohort 1) | Part B: Miransertib PS (Cohort 2) | Part B: Miransertib PROS/PS (Cohort 3) | Part B:Miransertib Compassionate Use/Expanded Access(Cohort 4)
Number analyzed (Participants) | 17 | 22 | 1 | 8 | 1
Participants | 2 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 48 months
Description: All-cause mortality was reported on all enrolled participants. Non-serious and serious AEs were reported on all participants who received at least one dose of study treatment. Per protocol, disease progression (DP) was not considered an AE unless related to treatment.
Arm/Group | Part A: Miransertib PROS/PS | Part B: Miransertib PROS (Cohort 1) | Part B: Miransertib PS (Cohort 2) | Part B: Miransertib PROS/PS (Cohort 3) | Part B: Miransertib Compassionate Use/Expanded Access (Cohort 4)
All-Cause Mortality (participants affected / at risk) | 1/17 | 0/22 | 0/1 | 0/8 | 0/2
Serious Adverse Events (participants affected / at risk) | 4/17 | 3/22 | 0/1 | 1/8 | 0/1
Other Adverse Events (participants affected / at risk) | 17/17 | 18/22 | 0/1 | 6/8 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Miransertib PROS/PS (N=17) | Part B: Miransertib PROS (Cohort 1) (N=22) | Part B: Miransertib PS (Cohort 2) (N=1) | Part B: Miransertib PROS/PS (Cohort 3) (N=8) | Part B: Miransertib Compassionate Use/Expanded Access (Cohort 4) (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Miransertib PROS/PS (N=17) | Part B: Miransertib PROS (Cohort 1) (N=22) | Part B: Miransertib PS (Cohort 2) (N=1) | Part B: Miransertib PROS/PS (Cohort 3) (N=8) | Part B: Miransertib Compassionate Use/Expanded Access (Cohort 4) (N=1)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 1 (3) | 0 (0) | 2 (6) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema of eyelid (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (11) | 2 (5) | 0 (0) | 4 (7) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (20) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (12) | 2 (3) | 0 (0) | 4 (10) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (6) | 0 (0) | 3 (7) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (4) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salivary duct obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 4 (6) | 0 (0) | 1 (3) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (24) | 5 (13) | 0 (0) | 2 (6) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fatigue (General disorders) | 2 (7) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lithiasis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Mucosal inflammation (General disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 15 (74) | 3 (3) | 0 (0) | 2 (8) | 0 (0)
Suprapubic pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 4 (10) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coxsackie viral infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scarlet fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (6) | 7 (13) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Viraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Anion gap (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood fibrinogen increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood insulin increased (Investigations) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 4 (6) | 0 (0)
Bone density decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibrin D dimer decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematocrit increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (8) | 1 (1) | 0 (0) | 4 (10) | 0 (0)
Lymphocyte count increased (Investigations) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Monocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (17) | 1 (2) | 0 (0) | 3 (5) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Platelet count decreased (Investigations) | 3 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 2 (4) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urine ketone body present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
White blood cell count decreased (Investigations) | 2 (3) | 1 (1) | 0 (0) | 2 (5) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (5) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperinsulinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (4) | 2 (5) | 0 (0) | 1 (2) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (14) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (27) | 2 (4) | 0 (0) | 3 (3) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (3) | 3 (5) | 0 (0) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 3 (9) | 2 (3) | 0 (0) | 2 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enuresis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perineal erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Testicular oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (17) | 3 (4) | 0 (0) | 2 (4) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (7) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (6) | 3 (3) | 0 (0) | 1 (4) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (3) | 0 (0) | 2 (2) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bullous haemorrhagic dermatosis (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphorrhoea (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Venous haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination due to business reasons

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to publish the results performed under this protocol, provided that such publication does not disclose any Confidential Information or trade secrets of the Sponsor (other than the data). The investigator agrees not to independently publish the findings except as part of an overall multicenter publication, unless approved in writing by the Sponsor or unless more than 12 months have elapsed since the last participant in the study has completed study treatment.

DOCUMENTS (2):
  • Study Protocol (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT03094832/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/32/NCT03094832/SAP_001.pdf